CLINICAL TRIAL: NCT02681406
Title: Impact of Enhancements to Smartphone Based Continuing Care for Alcohol Dependence
Brief Title: Smartphone Based Continuing Care for Alcohol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 819881
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment as Usual (No Intervention): Participants randomized to this condition will continue their schedules and treatments as they had been and just come in to see research staff for research visits.
- Telephone Monitoring and Counseling (Experimental): TMC - participants receive brief (20 minute) telephone counseling once weekly, then biweekly, etc for 12 months.
  Interventions: Behavioral: TMC
- ACHESS (Experimental): Participants are signed up for an addiction based smart phone application that connects them in an anonymous fashion to a social network of other people in the study who are also struggling with alcohol addiction and sober living.
  Interventions: Behavioral: ACHESS
- TMC + ACHESS (Experimental): Participants in this arm receive both interventions - the telephone counseling plus the ACHESS phone application.
  Interventions: Behavioral: ACHESS; Behavioral: TMC

INTERVENTIONS:
Behavioral: ACHESS — Smartphone based additions focused application, encouraging social support
  Arms: ACHESS; TMC + ACHESS
Behavioral: TMC — Brief telephone monitoring and counseling
  Arms: TMC + ACHESS; Telephone Monitoring and Counseling

SUMMARY:
Investigators will recruit 280 alcohol dependent patients in treatment programs in the Philadelphia area to test the efficacy and cost efficiency of a smartphone based application for treating alcohol addiction (ACHESS) with telephone monitoring and counseling (TMAC). Participation in the study lasts for 18 months with research visits at baseline, 3 months, 6 months, 9 months, 12 months, and 18 months. The intervention lasts 12 months.

DETAILED DESCRIPTION:
Continuing care is believed to be important in the effective management of patients with alcohol use disorders. New smartphone technology provides a novel way to provide personalized continuing care support. Dr. Gustafson and colleagues at the University of Wisconsin have developed an addiction version of CHESS (ACHESS), an automated smart phone system that provides a range of functions designed to directly support patients. In a recently completed NIAAA-funded continuing care study, ACHESS produced better drinking outcomes with alcoholics than treatment as usual.

The Principal Investigator of the current study, Dr. Jim McKay, and his colleagues at the Center of Continuum of Care in the Addictions have also developed a telephone-based approach to continuing care, Telephone Monitoring and Counseling (TMC), which has demonstrated efficacy in two randomized trials with alcohol-dependent patients. The TMC intervention is delivered through telephone contacts between patients and counselors, and makes use of information obtained in a brief assessment at the beginning of each call to determine the content of the session and to trigger adaptive changes in level of care over time.

Although both ACHESS and TMC use telephone technology, they have complementary strengths. ACHESS provides a range of automated 24/7 recovery support services, but does not include contact with a counselor. TMC, on the other hand, provides regular and sustained contact with the same counselor, but does not provide support between calls. The future of continuing care for alcohol use disorders is likely to involve both automated mobile technology and counselor contact, but little is known about how best to integrate these services.

To address this question, the study will feature a 2 x 2 design [ACHESS for 12 months (yes/no) x TMC for 12 months (yes/no)]. With this design, we will determine whether adding TMC to ACHESS produces superior outcomes to those obtained with TMC or ACHESS alone. This design will also enable replication of prior findings, and will provide the first direct comparison of TMC only vs. ACHESS only. In addition, economic analyses will be completed to determine the cost and cost-effectiveness of each intervention and their combination. The participants will be randomly assigned into one of the four conditions and followed for 18 months. The follow-ups will be at 3, 6, 9, 12, and 18 months post-baseline.

The subjects will be 280 patients diagnosed with alcohol abuse who are in a substance abuse treatment center in the Philadelphia area.

The risks of the research are conceived to be minimal (e.g., possible embarrassment) and consist of those incurred in providing self-report data on alcohol and drug-related history and social and psychiatric problems. There are minimal medical risks associated with research participation. There will be some risk of loss of confidentiality since the name, addresses and phone numbers of three contact people will be recorded by the staff for subject tracking purposes. However, all identifiable information will remain in a locked filling cabinet only accessible by the principle investigator and study staff. No identifying information will be programmed into the phone by the counselor. Although the participant is able to program numbers into the smartphone once they receive one, the counselor will review several measures for protecting the subjects' privacy, including password and pattern locks. All subjects will receive at a minimum treatment as usual in the programs from which they will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* have a DSM-V diagnosis of current, moderate to severe alcohol use disorder
* have completed 3 weeks of IOP
* be 18-75 years of age
* be able to provide the name and verified telephone number of at least two contacts to help reach participants for follow up appointments
* functionally literate and have sufficient ability to read a smart phone
* be willing to be randomized as part of the clinical trial

Exclusion Criteria:

* have a current psychotic disorder or dementia severe enough to prevent participation in treatment
* have an acute medical problem requiring immediate inpatient treatment
* are participating in other forms of treatment for substance abuse, besides IOP
* are unable to read/comprehend for informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-09; Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. McKay, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKay JR, Gustafson DH, Ivey M, Pe-Romashko K, Curtis B, Thomas T, Oslin DW, Polsky D, Quanbeck A, Lynch KG. Efficacy and comparative effectiveness of telephone and smartphone remote continuing care interventions for alcohol use disorder: a randomized controlled trial. Addiction. 2022 May;117(5):1326-1337. doi: 10.1111/add.15771. Epub 2021 Dec 23. PMID 34859519
- [Derived] McKay JR, Gustafson DH, Ivey M, McTavish F, Pe-Romashko K, Curtis B, Oslin DA, Polsky D, Quanbeck A, Lynch KG. Effects of automated smartphone mobile recovery support and telephone continuing care in the treatment of alcohol use disorder: study protocol for a randomized controlled trial. Trials. 2018 Jan 30;19(1):82. doi: 10.1186/s13063-018-2466-1. PMID 29382367

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual | Telephone Monitoring and Counseling | ACHESS | TMC + ACHESS
Started | 65 | 59 | 68 | 70
Completed | 49 | 35 | 42 | 58
Not Completed | 16 | 24 | 26 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Telephone Monitoring and Counseling | ACHESS | TMC + ACHESS | Total
Number analyzed (Participants) | 65 | 59 | 68 | 70 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.70 (9.93) | 46.07 (10.15) | 48.00 (9.21) | 46.72 (11.03) | 46.87 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 15 | 21 | 76
  Male | 44 | 40 | 53 | 49 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 3 | 3
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 53 | 49 | 59 | 55 | 216
  White | 9 | 8 | 6 | 8 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 65 | 59 | 68 | 70 | 262
Short Index of Problems - Revised (SIP-R [Mean (Standard Deviation); unit: units on a scale] — Alcohol Short Index of Problems 15 items Five subscales and total score. Total score (sum of items) is reported. Higher scores indicate worse outcome. Lowest possible score = 0; Highest possible score = 45
  units on a scale | 11.35 (3.88) | 11.47 (3.69) | 11.96 (4.00) | 12.36 (3.43) | 11.79 (3.75)
Timeline Follow Back [Mean (Standard Deviation); unit: percent days of heavy drinking] — Baseline Timeline Follow Back is a measure used to record daily use amounts, and goes back 90 days. We interview the study participants using calendars with anchors on them such as holidays or days important to the participant (mother's birthday) or to the region (a big local sports team win), to help them orient themselves and come up with their best informed responses to how many standard drinks they had that day. Percent days heavy drinking is the percent of the days we have data on, that were spent drinking heavily (5 or more for men; 4 or more for women).
  percent days of heavy drinking | 41.35 (29.40) | 45.34 (28.52) | 46.36 (28.59) | 46.86 (30.45) | 44.98 (29.24)

OUTCOME MEASURES:

1. Primary Outcome: Time Line Follow Back, Percent Heavy Alcohol Use
Description: The primary outcome measure will be percent days of heavy alcohol use (i.e., > 5 drinks/day for men, > 4 drinks/day for women) within each follow-up period. Studies have consistently supported the reliability and validity of the TLFB with alcohol dependent individuals. Frequency of heavy alcohol use was selected because alcohol-related problems are correlated with the frequency of heavy drinking days. This outcome is also sensitive to reductions in problematic or high risk use, which are particularly important in a disease management model.
Time Frame: 18 month: months 13 - 18 post baseline
Measure: Mean (Standard Error); unit: percentage of days heavy drinking
Arm/Group | Treatment as Usual | Telephone Monitoring and Counseling | ACHESS | TMC + ACHESS
Number analyzed (Participants) | 49 | 35 | 42 | 51
percentage of days heavy drinking | 8.10 (2.74) | 9.97 (3.33) | 8.79 (3.76) | 5.49 (1.79)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Treatment as Usual | Telephone Monitoring and Counseling | ACHESS | TMC + ACHESS
All-Cause Mortality (participants affected / at risk) | 0/65 | 2/59 | 3/68 | 1/70
Serious Adverse Events (participants affected / at risk) | 6/65 | 8/59 | 9/68 | 11/70
Other Adverse Events (participants affected / at risk) | 0/65 | 0/59 | 0/68 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (N=65) | Telephone Monitoring and Counseling (N=59) | ACHESS (N=68) | TMC + ACHESS (N=70)
Overdose hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
seizure disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Heart issues (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
diabetes (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
psychiatric problems (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Intestinal upset (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
kidney problems (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hysterectomy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cyst removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hand surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02681406/Prot_SAP_000.pdf